CLINICAL TRIAL: NCT04038606
Title: Quality of Life and Breast Cancer in Older Women
Brief Title: SEINIOR:Quality of Life and Breast Cancer in Older Women
Acronym: SEINIOR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Hospital Saint Quentin (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016-A00286-45
Record Dates: First submitted 2016-09-28; First posted 2019-07-31 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants completed a questionnaires that included the test sociodemographic characteristics and a number of standardized validated instruments translated in French language designed to assess for quality of life and psychological profile.
  Participants will undergo blood test, electrocardiogram, blood pressure monitoring, geriatric standard evaluation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- acceptance of mastectomy (Active Comparator): Assess the determinants of acceptance of mastectomy based on personal background,Measured by questionnaires: self-image (Rosenberg),personal background (level of fragility, self-image),quality of life SF-36, QLQC30,pain (BPI-SF) and Big Five Inventory.
  Interventions: Other: Determination of acceptance and / or rejection of mastectomy
- rejection of mastectomy (Experimental): Assess the determinants of rejection of mastectomy based on personal background, Measured by questionnaires: self-image (Rosenberg),personal background (level of fragility, self-image),quality of life SF-36, QLQC30,pain (BPI-SF) and Big Five Inventory.
  Interventions: Other: Determination of acceptance and / or rejection of mastectomy

INTERVENTIONS:
Other: Determination of acceptance and / or rejection of mastectomy — Blood exams,Participants completed a questionnaire translated in French language : Rosenberg,SF-36, QLQC30, Big Five Inventory,BPI-SF.:-)

SUMMARY:
Background :

Breast cancer is a disease that occurs primarily in elderly women: 54057 of breast cancer occurred on women in 2008, 15.2% were between 75 and 84 years and 5.4% were over 85 years. Elderly women cancers care exposes to several problems: the opportunity for screening, knowing that mammography is not recommended after 75 years old, and the level of treatment depending on the background and the existence of weaknesses. It should determine whether patients are in adequate physiological condition to tolerate classical and "complete" treatment or conversely in a precarious state with advanced fragility, justifying only lightened and adapted symptomatic treatment.

Purpose :

The purpose of this research theme is to assess the quality of life of elderly patients who underwent mastectomy for breast cancer. The objectives are:

* Assess the determinants of acceptance and / or rejection of mastectomy based on personal background (level of fragility, self-image) and linked to cancer
* Assess the quality of life, 6 months later, of women who underwent or not mastectomy, and appreciate the determinants

Abstract :

The total mastectomy allow, oncologically, a more valid treatment than a lumpectomy, in many cases of women suffering from a breast cancer, but its relevance and acceptability are poorly known. Some think that an elderly woman, postmenopausal, is less concerned with her aesthetics and feminine attributes, which would allow her to accept easily the mastectomy.

The research hypothesis is that the acceptability of mastectomy is not good in elderly women

DETAILED DESCRIPTION:
Primary outcome:

Better detection of comorbidity and geriatric syndromes in vulnerable patients Better detection of a degradation of the quality of life at D0 (at diagnosis)

Secondary outcomes:

Better support for quality of life and psychological support after mastectomy (revaluation to 6 months) Integration of patients in the geriatric sector and implementation of regular monitoring Study design: prospective, multicenter

ELIGIBILITY:
Inclusion Criteria:

1. Elderly patients about or over 75 years
2. Female
3. Patients in whom a diagnosis of breast cancer with surgical indication for mastectomy with or without lymph node dissection is discussed
4. Ability to understand and give freely consent
5. Informed consent signed
6. Patient affiliated to the social security or entitled

Exclusion Criteria:

1. Patients under 75 years
2. Male
3. Patients under legal protection

Ages: 75 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2016-12-15 (Actual); Primary Completion 2020-12-15 (Estimated); Study Completion 2020-12-15 (Estimated)

PRIMARY OUTCOMES:
Evaluation of quality of life change by SF-36 (The Short Form Health Survey) between baseline and six months | Baseline and 6 months
  the 36-Item Short Form Health Survey (SF-36). SF-36 is a set of generic, coherent, and easily administered quality-of-life measures. These measures rely upon patient self-reporting and are now widely utilized monitoring and assessment of care outcomes in adult patients.
  a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability

SECONDARY OUTCOMES:
QLQ-C30 (Global Health Status) | Baseline and 6 months
  Quality of life (QoL or QOL) is the perceived quality of an individual's daily life, that is, an assessment of their well-being or lack thereof. This includes all emotional, social and physical aspects of the individual's life;All of the scales and single-item measures range in score from 0 to 100.
Psychological profile | Baseline and 6 months
  Big Five Inventory (BFI),personality inventory for research settings, minimum = 45 points and maximum scores = 180 points .

CONTACTS AND LOCATIONS:
Overall Officials: ATTIER-ZMUDKA Dr Jadwiga, PI, Principal Investigator — Saint Quentin Hospital
Locations (1):
- Centre Hospitalier de Saint-Quentin;, Saint-Quentin, Aisne, France

IPD SHARING:
Plan to Share IPD: No
Participants completed a questionnaire that included the test sociodemographic characteristics and a number of standardized validated instruments translated in French language designed to assess for quality of life and psychological profile.
  Participants will undergo blood test, electrocardiogram, blood pressure monitoring, geriatric standard evaluation.